CLINICAL TRIAL: NCT03362580
Title: Prevalence and Risk Factors of Epiretinal Membrane in Diabetic and Non-diabetic Patients: a Prospective, Cross-sectional and Comparative Study
Brief Title: Prevalence and Risk Factors of Epiretinal Membrane in Diabetic and Non-diabetic Patients
Status: Completed | Type: Observational
Sponsor: Laurence Postelmans (Other)
Responsible Party: Sponsor-Investigator, Laurence Postelmans, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-ERM
Record Dates: First submitted 2017-11-16; First posted 2017-12-05 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Epiretinal Membrane
Keywords: Epiretinal Membrane; Diabetes
MeSH Terms: conditions — Epiretinal Membrane; Diabetes Mellitus | interventions — Slit Lamp Microscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients diagnosed with diabetes mellitus, type 1 or type 2, aged 15 years or older
  Interventions: Device: Slit lamp examination; Device: Undilated 7-field color fundus photography; Device: Color scan; Device: Spectral domain optical coherence tomography
- Group B: Patients non-diagnosed with diabetes mellitus, aged 15 years or older
  Interventions: Device: Slit lamp examination; Device: Undilated 7-field color fundus photography; Device: Color scan; Device: Spectral domain optical coherence tomography

INTERVENTIONS:
Device: Slit lamp examination — The slit lamp is an instrument consisting of a high-intensity light source that can be focused to shine a thin sheet of light into the eye.Examination performed without pupil dilatation.
Device: Undilated 7-field color fundus photography — Undilated 7-field color fundus photography with Cobra fundus camera. The examination will be done without pupil dilatation; but in case of very small pupils one drop of tropicamide will be instilled, after anterior segment observation with the slit lamp. Two ophthalmologists will assess fundus photos and OCT (Spectral domain optical coherence tomography) frames, to determine whether or not an ERM is present.
Device: Color scan — Multicolor photo. The examination will be done without pupil dilatation; but in case of very small pupils one drop of tropicamide will be instilled, after anterior segment observation with the slit lamp.
Device: Spectral domain optical coherence tomography — Spectral domain optical coherence tomography (OCT) with Heidelberg Retina Tomography device. The examination will be done without pupil dilatation; but in case of very small pupils one drop of tropicamide will be instilled, after anterior segment observation with the slit lamp.Two ophthalmologists will assess fundus photos and OCT frames, to determine whether or not an ERM is present.

SUMMARY:
Numerous terms have been used to describe epiretinal membrane (ERM): macular pucker, epimacular membrane, surface-wrinkling retinopathy, cellophane maculopathy and preretinal macular fibrosis. It is, by definition, a fibrocellular tissue found on the inner surface of the retina. It is semi-translucent and proliferates on or above the surface of the internal limiting membrane. It causes blurring and metamorphopsia, while mild cases are often asymptomatic.

ERM presence can degrade the acuity and the quality of vision, thus affecting the quality of life. There is evidence that it also has an adverse impact to the treatment options for patients suffering from macular disorders. More specifically, regarding to diabetic retinopathy, ERM seems to have a bidirectional etiopathogenetic relationship with its course and complications.

The aim of this study is to know the prevalence of ERM in the Brussel's population, the risk factors predisposing to ERM formation and if diabetic patients have a significantly higher prevalence of ERM in comparison to general population.

ELIGIBILITY:
Inclusion Criteria:

-Subjects examined in the general or diabetes screening consultations of the Ophthalmology Department of the CHU Brugmann Hospital

Exclusion Criteria:

* Women pregnant or breast-feeding
* Hypersensitivity to tropicamide
* Any macular pathology other than diabetic maculopathy
* Prior retinal photocoagulation
* Prior intravitreal injection
* Prior retinal surgery

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects examined in the general or diabetes screening consultations of the Ophtalmology Department of the CHU Brugmann Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Age | First standard of care consultation, up to 3 months
  Age
Gender | First standard of care consultation, up to 3 months
  Gender
Population sub-type | First standard of care consultation, up to 3 months
  Population sub-type: Caucasian, African, Asian, Indian, American or Other
Diabetes type (for group A) | First standard of care consultation, up to 3 months
  Diabetes type (for group A)
Diabetic Retinopathy classification | First standard of care consultation, up to 3 months
  Diabetic Retinopathy classification, if diagnosed (according to the Early Treatment of Diabetic Retinopathy Study (ETDRS) classification)
Duration of medical treatment of diabetes | First standard of care consultation, up to 3 months
  Duration of medical treatment of diabetes (measured in months)
HbA1C (Glycated Haemoglobin) rate | First standard of care consultation, up to 3 months
  HbA1C rate (according to recent blood test)
Smoking status | First standard of care consultation, up to 3 months
  Smoking status
Previous cataract surgery | First standard of care consultation, up to 3 months
  Previous cataract surgery
Diagnose of ERM | First standard of care consultation, up to 3 months
  Diagnose of ERM
Educational level | First standard of care consultation, up to 3 months
  Educational level

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Postelmans, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium